CLINICAL TRIAL: NCT03665194
Title: A Randomised, Double Blind, Placebo Controlled Phase I Study to Investigate the Effects of Systemically Absorbed Cortexolone 17α-propionate (and Its Metabolites) on QT Interval Following Repeat Topical Administration in Healthy Volunteers
Brief Title: A Study to Investigate the Effects of Cortexolone 17α-propionate (and Its Metabolites) on Healthy Volunteers' Heart
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cassiopea SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CB-03-01/33
Record Dates: First submitted 2018-06-18; First posted 2018-09-11 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Healthy Volunteers
Keywords: QT/QTc Interval

STUDY DESIGN:
Intervention Model Description: Thirty-two volunteers will be enrolled and evaluated (i.e. complete the study). Subjects will be dosed in four groups of eight (purely for logistical reasons relating to the procedure times expected with dosing and ECG). Volunteers will receive either the active drug or matching placebo in a 3:1 ratio. Therefore within each cohort, six volunteers will receive the active drug and two will receive matching placebo.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cortexolone 17α-propionate 7.5% solution (Experimental)
  Interventions: Drug: Cortexolone 17α-propionate solution
- Vehicle solution (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cortexolone 17α-propionate solution — Single topical application to be applied twice daily (0 hour and 12 hour) on Days 1-3 and Once Daily (0 hour) on Day 4.
  Arms: Cortexolone 17α-propionate 7.5% solution
Drug: Placebo — matching placebo
  Arms: Vehicle solution

SUMMARY:
This is a randomised, double blind placebo controlled Phase I study which will assess the safety, tolerability and PK of Cortexolone 17α-propionate (and its metabolites), and its effects on the QTc interval when administered as multiple doses to healthy adult volunteers. Volunteers will receive a morning and evening dose (12 hours apart) of 225 mg (3 mL Cortexolone 17α-propionate applied topically as a 7.5 % solution (75 mg in 1 mL), giving a total daily dose of 450 mg (6 mL) per individual.

DETAILED DESCRIPTION:
Thirty-two volunteers will be enrolled and evaluated (i.e. complete the study). Subjects will be dosed in four groups of eight (purely for logistical reasons relating to the procedure times expected with dosing and ECG). Volunteers will receive either the active drug or matching placebo in a 3:1 ratio. Therefore within each cohort, six volunteers will receive the active drug and two will receive matching placebo.

Volunteers will be screened within 20 days prior to entering the study on Day -1. Each volunteer will receive verbal and written information followed by signing of the ICF prior to any screening procedures taking place. Volunteers will be admitted to the study unit on Day -1, dosed twice daily on Days 1-3 and once on Day 4 (morning dose only). They will be discharged on Day 6 and will have a telephone follow-up on Day 14. If they report any relevant Adverse Event (AE) they will be invited to attend the unit for an outpatient visit as close to Day 14 as is possible.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥18 and ≤40 years at the date of signing informed consent which is defined as the beginning of the Screening Period.
2. Subjects must have a body mass index (BMI) between 18.0-25.0 kg/m² inclusive.
3. Subjects must be bald, have a shaved head, or be willing to have their head shaved.
4. Female subjects who are either: (a) Non-childbearing potential, e.g. post-menopausal (as defined as amenorrhoea for at least 12 months with no alternative medical cause) or permanently sterile (permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy) OR (b) Childbearing potential AND (if heterosexually active) agree to use at least one form of highly effective contraception as defined below, starting at least one menstrual cycle before first study drug administration and continuing until at least 3 months after the end of the systemic exposure of the study drug.

   Highly effective contraceptive methods for females are as follows:
   * Combined (oestrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation as follows:

     * Oral
     * Intravaginal
     * Transdermal
   * Progestogen-only hormonal contraception associated with inhibition of ovulation as follows: o Oral

     * Injectable
     * Implantable
   * Intrauterine device (IUD)
   * Intrauterine hormone-releasing system (IUS)
   * Bilateral tubal occlusion
   * Male partner vasectomised (with documented evidence of azoospermia if possible)
5. Male subjects, if heterosexually active and with a female partner of childbearing potential or a pregnant or breastfeeding partner, must agree to use barrier contraception (male condom) for the treatment period and for at least three months after the end of the systemic exposure of the study drug. Female partners of male subjects who are of childbearing potential must use one or more forms of highly effective contraception as defined above, starting at least one menstrual cycle before (their male subject's) first study drug administration and continuing until at least three months after the end of their male partner's systemic exposure to the study drug.

   For male subjects who have had a vasectomy (with documented evidence of azoospermia if possible) and agree to use a barrier method (male condom) for the stated time period, no additional contraceptive method is required by their female partner.
6. Subjects must agree not to donate sperm or ova from the time of the first administration of study medication until 3 months after the end of the systemic exposure of the study drug.
7. Satisfactory medical assessment with no clinically significant or relevant abnormalities as determined by medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory evaluation (haematology, biochemistry, coagulation and urinalysis) that is reasonably likely to interfere with the subject's participation in or ability to complete the study as assessed by the investigator.
8. Ability to provide written, personally signed, and dated informed consent to participate in the study, in accordance with the ICH Good Clinical Practice (GCP) Guideline E6 (1996) and applicable regulations, before completing any study-related procedures.
9. An understanding, ability, and willingness to fully comply with study procedures and restrictions.

Exclusion Criteria:

1. Current or recurrent disease (e.g., cardiovascular, haematological, neurological, endocrine, renal, liver, gastrointestinal, hepatic or other conditions) that could affect the action, absorption, or disposition of Cortexolone 17α-propionate, or could affect clinical assessments or clinical laboratory evaluations.
2. Current or relevant history of any physical or psychiatric illness that may require treatment or make the subject unlikely to fully comply with the requirements of the study or complete the study, or any condition that presents undue risk from the investigational product or study procedures.
3. Any other significant disease or disorder which, in the opinion of the investigator, may put the subject at unacceptable risk because of participation in the study, may influence the result of the study, or may affect the subject's ability to participate in the study.
4. History of any pathology affecting the skin such as eczema, psoriasis or any skin hypersensitivity.
5. Have tattoos on the scalp or thigh which would affect the area for topical application of the trial drug.
6. The history or presence of any of the following cardiac conditions: known structural cardiac abnormalities; family history of long QT syndrome; cardiac syncope or recurrent, idiopathic syncope; exercise related clinically significant cardiac events.
7. Any clinically significant abnormalities in rhythm, conduction or morphology of resting ECG or clinically important abnormalities that may interfere with the interpretation of QTc interval changes. This includes subjects with any of the following (at screening, Day -1 or pre-dose of Day 1):

   * Sinus node dysfunction.
   * Clinically significant PR (PQ) interval prolongation.
   * Intermittent second or third degree AV block.
   * Complete bundle branch block.
   * Sustained cardiac arrhythmia's including (but not limited to) atrial fibrillation or supraventricular tachycardia; any symptomatic arrhythmia with the exception of isolated extra systoles.
   * More than 200 ventricular ectopic beats in 24 hours.
   * Ventricular tachycardia (ventricular tachycardia defined as ≥ 3 successive ventricular ectopic beats at a rate of > 120 bpm).
   * Abnormal T wave morphology.
   * QT interval corrected using the Fridericia's formula (QTcF) > 450 ms.
   * Any other ECG abnormalities in the standard 12-lead ECG and 24-hour 12 lead Holter ECG or an equivalent assessment which in the opinion of the investigator will interfere with the ECG analysis.

   Subjects with borderline abnormalities may be included if the deviations do not pose a safety risk, and if agreed between the appointed Cardiologist and the investigator.
8. Has vital signs outside of the following normal range at screening, Day -1 or Day 1 predose:

   1. Blood pressure (BP):

      Supine BP (after at least 5 minutes of supine rest):
      * Systolic blood pressure: 90 - 140 mmHg.
      * Diastolic blood pressure: 40 - 90 mmHg.
   2. Supine pulse rate after at least 5 minutes of rest: 45 - 100 bpm .
9. Positive test for Hepatitis B surface antigen (HBsAg), Hepatitis C antibody (HCV Ab), or human immunodeficiency virus antibody (HIV Ab) at screening;
10. Subjects who are pregnant, breast feeding or lactating.
11. Any clinically relevant abnormal laboratory results (including hepatic and renal panels, complete blood count, chemistry panel, coagulation and urinalysis), and vital signs, or physical findings at screening, pre-dose of Day 1 (as judged by the investigator). In case of uncertain or questionable results, tests performed during screening may be repeated before randomization to confirm eligibility or judged to be clinically irrelevant for healthy subjects.
12. Positive test results for alcohol or drugs of abuse at screening or Day -1.
13. Presence or history of drug or alcohol abuse in the last 5 years, or the inability to refrain from alcohol use from 48 hours before screening, dosing and each scheduled visit until the end of the study. Alcohol abuse is defined as regular weekly intake of more than 14 units, using the following NHS alcohol tracker http://www.nhs.uk/Tools/Pages/drinks-tracker.aspx.
14. Use of tobacco in any form (e.g., smoking or chewing) or other nicotine-containing products in any form (e.g., gum, patch, electronic cigarettes) within 3 months prior to the planned first day of dosing.
15. Use of prescription medications within 14 days or 10 half-lives (whichever is longer) prior to Day 1 of the dosing period, or any over-the-counter (OTC) medication (including multivitamin, herbal, or homeopathic preparations, excluding hormonal contraception, hormone-replacement therapy, and/or an occasional dose of acetaminophen) within 7 days prior to Day 1 of the dosing period.
16. Consumption of herbal remedies or dietary supplements containing St. John's Wort in the three weeks before the planned Day 1 of the dosing period.
17. Consumption of drugs or other substances known to be potent inhibitors or inducers of CYP P450s in the three weeks before the planned Day 1 of the dosing period. This includes food or drink products containing cranberry, pomegranate, star fruit, grapefruit, pomelos, exotic citrus fruits or Seville oranges (including marmalade and juices made from these fruits).
18. Consumption of caffeine, caffeine-containing or xanthine-containing products, energy drinks containing taurine or glucuronolactone within 48 hours prior to the planned first study drug administration.
19. Has received an investigational product or been treated with an investigational device within 90 days prior to first drug administration and will not start any other investigational product or device study within 90 days after last study drug administration.
20. Known or suspected intolerance or hypersensitivity to the investigational product, any closely related compound or any of the stated ingredients.
21. History of significant allergic reaction (anaphylaxis, angioedema) to any product (food, pharmaceutical, etc).
22. Has donated or lost 400 mL blood or more within the last 16 weeks preceding the first day of dosing.
23. Has a mental incapacity or language barriers precluding adequate understanding, co-operation, and compliance with the study requirements.

    Cassiopea S.p.A. CONFIDENTIAL 30 April 2018 Protocol Ref: CB-03-01/33 Final Version 5.0 Page 30 of 43 RPL Study No. C16021 C16021_Protocol_v5.0_30Apr2018
24. An inability to follow a standardized diet and meal schedule or inability to fast, as required during the study.
25. Prior screen failure (where the cause of the screen failure is not deemed to be temporary), randomization, participation, or enrolment in this study. Subjects who initially failed due to temporary non-medically significant issues are eligible for re-screening once the cause has resolved.
26. Objection by the General Practitioner (GP) to the subject entering the study.
27. Subjects with any medical history, conditions, or risks that, in the opinion of the investigator, may interfere with the subject's full participation in the study or compliance with the protocol, or may pose any additional risk for the subject or confound the assessment of the subject or outcome of the study.

    -

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-06-06 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-09-12 (Actual)

PRIMARY OUTCOMES:
PK parameters of Cortexolone 17α-propionate and the two main metabolites Cortexolone 21-propionate (M1) and Cortexolone (M2) | Samples will be collected 1hour pre IMP administration and at 2, 3, 4, 5, 6, 7, 8, 9, 10,12 hours post IMP administration on Day1 and Day4. Further samples will be collected at 24 hours (Day 5) and 48 hours (Day 6) after the final dose on Day 4.
  Cmax: Maximum observed plasma concentration Days 1 and 4
PK parameters of Cortexolone 17α-propionate and the two main metabolites Cortexolone 21-propionate (M1) and Cortexolone (M2) | Samples will be collected 1hour pre IMP administration and at 2, 3, 4, 5, 6, 7, 8, 9, 10,12 hours post IMP administration on Day1 and Day4. Further samples will be collected at 24 hours (Day 5) and 48 hours (Day 6) after the final dose on Day 4.
  tmax: Time of maximum observed plasma concentration
PK parameters of Cortexolone 17α-propionate and the two main metabolites Cortexolone 21-propionate (M1) and Cortexolone (M2) | Samples will be collected 1hour pre IMP administration and at 2, 3, 4, 5, 6, 7, 8, 9, 10,12 hours post IMP administration on Day1 and Day4. Further samples will be collected at 24 hours (Day 5) and 48 hours (Day 6) after the final dose on Day 4.
  t½: Apparent plasma terminal elimination half-life
PK parameters of Cortexolone 17α-propionate and the two main metabolites Cortexolone 21-propionate (M1) and Cortexolone (M2) | Samples will be collected 1hour pre IMP administration and at 2, 3, 4, 5, 6, 7, 8, 9, 10,12 hours post IMP administration on Day1 and Day4. Further samples will be collected at 24 hours (Day 5) and 48 hours (Day 6) after the final dose on Day 4.
  AUC0-24h: Area under the plasma concentration-time curve from time zero to 24 hours, calculated by the linear/log trapezoidal rule
PK parameters of Cortexolone 17α-propionate and the two main metabolites Cortexolone 21-propionate (M1) and Cortexolone (M2) | Samples will be collected 1hour pre IMP administration and at 2, 3, 4, 5, 6, 7, 8, 9, 10,12 hours post IMP administration on Day1 and Day4. Further samples will be collected at 24 hours (Day 5) and 48 hours (Day 6) after the final dose on Day 4.
  AUC0-t: Area under the plasma concentration-time curve from time zero up to the last quantifiable concentration
PK parameters of Cortexolone 17α-propionate and the two main metabolites Cortexolone 21-propionate (M1) and Cortexolone (M2) | Samples will be collected 1hour pre IMP administration and at 2, 3, 4, 5, 6, 7, 8, 9, 10,12 hours post IMP administration on Day1 and Day4. Further samples will be collected at 24 hours (Day 5) and 48 hours (Day 6) after the final dose on Day 4.
  AUC0-inf: Area under the plasma concentration-time curve from time zero to infinity
PK parameters of Cortexolone 17α-propionate and the two main metabolites Cortexolone 21-propionate (M1) and Cortexolone (M2) | Samples will be collected 1hour pre IMP administration and at 2, 3, 4, 5, 6, 7, 8, 9, 10,12 hours post IMP administration on Day1 and Day4. Further samples will be collected at 24 hours (Day 5) and 48 hours (Day 6) after the final dose on Day 4.
  CL: Blood clearance
PK parameters of Cortexolone 17α-propionate and the two main metabolites Cortexolone 21-propionate (M1) and Cortexolone (M2) | Samples will be collected 1hour pre IMP administration and at 2, 3, 4, 5, 6, 7, 8, 9, 10,12 hours post IMP administration on Day1 and Day4. Further samples will be collected at 24 hours (Day 5) and 48 hours (Day 6) after the final dose on Day 4.
  λz: Terminal elimination rate constant
PK parameters of Cortexolone 17α-propionate and the two main metabolites Cortexolone 21-propionate (M1) and Cortexolone (M2) | Samples will be collected 1hour pre IMP administration and at 2, 3, 4, 5, 6, 7, 8, 9, 10,12 hours post IMP administration on Day1 and Day4. Further samples will be collected at 24 hours (Day 5) and 48 hours (Day 6) after the final dose on Day 4.
  CLr: Renal clearance
PK parameters of Cortexolone 17α-propionate and the two main metabolites Cortexolone 21-propionate (M1) and Cortexolone (M2) | Samples will be collected 1hour pre IMP administration and at 2, 3, 4, 5, 6, 7, 8, 9, 10,12 hours post IMP administration on Day1 and Day4. Further samples will be collected at 24 hours (Day 5) and 48 hours (Day 6) after the final dose on Day 4.
  Vz: Volume of distribution
PK parameters of Cortexolone 17α-propionate and the two main metabolites Cortexolone 21-propionate (M1) and Cortexolone (M2) | Samples will be collected 1hour pre IMP administration and at 2, 3, 4, 5, 6, 7, 8, 9, 10,12 hours post IMP administration on Day1 and Day4. Further samples will be collected at 24 hours (Day 5) and 48 hours (Day 6) after the final dose on Day 4.
  MRT: Mean residence time
QT interval changes | Day1 (each hour starting from 2 till 12 hours post IMP administration), Day 4 (each hour starting from 2 till 12 hours post IMP administration), Day 5 (24 hs post last IMP administration) and Day 6 (48 hs post last IMP administration).
  QT intervals will be assessed using triplicate 12-lead ECGs electronically recorded at each time point and evaluated by a blinded select cardiologist

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse event | Day1, 2, 3, 4, 5, 6 and 14
Proportion of subjects with skin reaction | Day1, 2, 3, 4, 5, 6 and 14 (if applicable)
  Skin reactions at the site of application will be assessed using a standardised in-house method. Any pain will be assessed using a Visual Analogue Scale (O-10).
Proportion of subjects with clinically significant changes in laboratory safety tests (haematology, chemistry, coagulation and urinalysis) | Haematology, chemistry and coagulation: Day-1/1, 3, 5 and 14. Urinalysis: Day-1 and Day 14
Proportion of subjects with abnormalities on electrocardiogram (ECG) | Day1, 4, 6 and 14
Proportion of subjects with clinically significant changes in vital signs (systolic blood pressure, diastolic blood pressure, pulse rate and temperature) | Day1, 2, 3, 4, 5 and 14

CONTACTS AND LOCATIONS:
Overall Officials: Jorg Taubel, MD FFPM, Principal Investigator — Richmond Pharmacology Limited
Locations (1):
- Richmond Pharmacology Ltd, London, United Kingdom